CLINICAL TRIAL: NCT02160197
Title: A Randomised Controlled Trial of Outcome of Different Post Operative Rehabilitation Regime Following Internally Fixed Ankle Fractures
Brief Title: Outcome of Rehabilitation Following Internally Fixed Ankle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Countess of Chester NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Wei Yee Leong, Clinical Research Registrar Trauma and Orthopaedic Surgery, Countess of Chester NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 142804
Record Dates: First submitted 2014-06-09; First posted 2014-06-10 (Estimated); Last update posted 2014-06-10 (Estimated); Status verified 2014-06

CONDITIONS: Ankle Fractures; Fracture
Keywords: Ankle Fractures; Fracture Fixation; Early Ambulation; Fracture Healing; Return to Work
MeSH Terms: conditions — Ankle Fractures; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Immobilisation (No Intervention): No immobilisation post op, allowing patients to weight bear as tolerated.
- Functional Bracing (Active Comparator): Immobilise patients in Functional brace, allowing patients to weight bear as tolerated.
  Interventions: Device: Aircast XP Walker boot
- Plaster Immobilisation (Active Comparator): Immobilise patients in plaster, allowing patients to weight bear as tolerated.
  Interventions: Device: Plaster Immobilisation

INTERVENTIONS:
Device: Aircast XP Walker boot — Ankle boot allowing weight bearing as tolerated
  Other Names: Functional Bracing
  Arms: Functional Bracing
Device: Plaster Immobilisation — Plaster immobilisation with no weight bearing allowed.
  Arms: Plaster Immobilisation

SUMMARY:
The purpose of this study is to examine the effect of variations in practice, ranging from early functional rehabilitation to complete immobilsation in post operative patients with ankle fixation following fractures. The primary goal of any post-operative regimen is to attain full weight-bearing and as close to pre-injury levels of activity as soon as possible.

We seek to establish the effect on (1) functional outcome, (2) complication rates and (3) time to return to work of three different approaches to rehabilitation after ankle fracture fixation in order to produce a standardised, evidence-based guideline for our unit. We also aim to perform a cost analysis for each approach.

DETAILED DESCRIPTION:
Although the indications for fixation of an ankle fracture are relatively clear, controversy exists with regards the post-operative management of these fractures.

This is a prospective randomised controlled trial. All patients admitted to the Countess of Chester NHS Foundation Trust Orthopaedic Unit for ankle fracture fixation who met the set study inclusion criteria will be given a patient information pack regarding the trial and asked to complete a consent form to enter the trial AFTER their operation has been performed. All patients will initially have their ankle immobilised in a below knee backslab applied in theatre and reviewed at 2 weeks in the plaster room for removal of plaster and sutures. At this setting the patient will be randomised to 1 of 3 rehabilitation arms using a sealed envelope technique. All patients data will be anonymised following generation of a randomisation number.

3 Orthopaedic Consultants (JH,KT,EW) will thereafter supervise follow-up of the study population until discharge at 1 year. Outcome measures recorded include patient -reported functional scores (MOxFQ); clinical assessment of range of motion, complication rates (loss of reduction); pain scores, satisfaction rates and return to work. Clinic review organised at 2 weeks for randomisation, 6 weeks for first post-op xrays and removal of plaster/ brace, 8 weeks for clinical review specifically range of movement achievable at ankle, 3 months with repeat Xray and clinical assessment, and final clinical review in clinic at 6 months in the fracture clinic. Telephone/ postal questionnaire to gather MoXFQ scores at 1 year.

There are no ethical or legal issues related to the studies.

One potential concern will be loss of reduction and fixation of ankle fractures following weight bearing without immobilisation. However, a study published by Gul et al in 2007 relating to immediate weight-bearing of operatively treated ankle fractures without immobilisation in cast showed no evidence of loss of reduction or hardware failure compared to historical controls.

Patients will be reviewed closely in the early period for loss of reduction as a safety outcome measure and the result will be monitored closely with earlier termination of trial should there be a concern. There will be monthly data review and monitoring during a research meeting.

Reference

Gul AG, Batra S, Meehmood S, Gillham N. Immediate unprotected weight-bearing of operatively treated ankle fractures. Acta Orthop Belgica 2007;73:360-365.

ELIGIBILITY:
Inclusion Criteria:

* Unstable and/or displaced Weber B ankle fractures
* Able to give informed consent and follow instructions
* Previously independently mobile without previous ankle surgery
* Closed isolated ankle injury
* Not known to be neuropathic or osteoporotic
* Treated with standard Small Frag AO technique ie. Lag screws plus 1/3 tubular plate for fibula fixation and 2 screws/TBW on medial side with wounds closed using 2.0 vicyl and nonabsorbable monofilament to skin. (Standard AO ankle fixation technique)

Exclusion Criteria:

* Weber C ankle fractures
* Patient from outside of region where follow-up will be in a different unit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
MOxFQ score (Manchester and Oxford Foot Questionaire | 1 year
  16-item Patient Reported Outcome (PRO) measures developed and validated for use in clinical trials involving foot surgery. These self-administered PROs assesses how foot problems impair health-related quality of life can be completed before and after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Y Leong, MBChB,MRCS, Principal Investigator — Countess of Chester NHS Foundation Trust
Locations (1):
- Countess of Chester NHS Foundation Trust, Chester, Cheshire, United Kingdom

REFERENCES:
- [Background] Gul A, Batra S, Mehmood S, Gillham N. Immediate unprotected weight-bearing of operatively treated ankle fractures. Acta Orthop Belg. 2007 Jun;73(3):360-5. PMID 17715727
- [Background] Egol KA, Dolan R, Koval KJ. Functional outcome of surgery for fractures of the ankle. A prospective, randomised comparison of management in a cast or a functional brace. J Bone Joint Surg Br. 2000 Mar;82(2):246-9. PMID 10755435
- [Background] van Laarhoven CJ, Meeuwis JD, van der WerkenC. Postoperative treatment of internally fixed ankle fractures: a prospective randomised study. J Bone Joint Surg Br. 1996 May;78(3):395-9. PMID 8636173